CLINICAL TRIAL: NCT03253055
Title: The Interrelationship Between Vitamin D, Bone, Illness, Injury and Its Impact on Exercise Performance
Brief Title: The D-BIICEP Study
Acronym: D-BIICEP
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Responsible Party: Principal Investigator, Saskia Wilson-Barnes, PhD Research Fellow, University of Surrey
Other Study IDs: D-BIICEP
Record Dates: First submitted 2017-08-08; First posted 2017-08-17 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Vitamin D Deficiency
Keywords: Physical Performance; Bone; Illness; Injury
MeSH Terms: conditions — Vitamin D Deficiency; Wounds and Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma and Serum samples obtained at baseline and visit 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Male Athletes: DEXA, pQCT, lifestyle questionnaire, muscular strength measurements, aerobic fitness, blood draw and finger prick test.
  Interventions: Radiation: DEXA; Radiation: pQCT; Other: Lifestyle Questionnaire; Other: Aerobic Fitness; Other: Muscular Strength; Biological: Blood draw and finger prick test; Other: Muscular Power
- Female Athletes: DEXA, pQCT, lifestyle questionnaire, muscular strength measurements, aerobic fitness, blood draw and finger prick test.
  Interventions: Radiation: DEXA; Radiation: pQCT; Other: Lifestyle Questionnaire; Other: Aerobic Fitness; Other: Muscular Strength; Biological: Blood draw and finger prick test; Other: Muscular Power
- Controls: DEXA, pQCT, lifestyle questionnaire, muscular strength measurements, aerobic fitness, blood draw and finger prick test.
  Interventions: Radiation: DEXA; Radiation: pQCT; Other: Lifestyle Questionnaire; Other: Aerobic Fitness; Other: Muscular Strength; Biological: Blood draw and finger prick test; Other: Muscular Power

INTERVENTIONS:
Radiation: DEXA — Dual energy X-ray absorptiometry (DEXA): a total of two scans will be performed, one for the assessment of whole body bone mineral density and body composition, and the other scan is performed to specifically assess fracture risk by scanning the hip and femoral head. Effective exposure doses for these scans are ~8uSv and ~4uSv respectively.
  Other Names: DXA
Radiation: pQCT — A total of one scan will be performed on the non-dominant Tibia, the effective exposure dose will be between 1.5-1.8uSV.
Other: Lifestyle Questionnaire — Participants are required to record their lifestyle, diet (5-day self reported), physical activity (IPAQ questionnaire), injury and illness incidence.
Other: Aerobic Fitness — Aerobic fitness will be tested using a VO2 max exercise protocol using a stationary cycle ergometer, the participants will be expected to perform this to maximal effort or exhaustion.
Other: Muscular Strength — Muscular strength of the knee extensor and handgrip muscles will be determined using an Isokinetic Dynamometer and a handgrip dynamometer respectively.
Biological: Blood draw and finger prick test — 15ml of whole blood will be collected for the measurement of fasting serum 25(OH)D levels, parathyroid hormone, C-terminal telopeptide (CTX) and full blood count
Other: Muscular Power — Muscular power will be determined using an optical measurement system consisting of a transmitting and receiving bar to determine jump height through the interpretation of jump flight of the participant (reported in cm). The equipment used is an Optojump.

SUMMARY:
Athletes and active individuals have been identified as an at-risk group for a low vitamin D status, specifically those residing in countries of higher latitude (such as the United Kingdom). This especially applies to those who train indoors for their sport, this is because Vitamin D is primarily produced following skin exposure to ultraviolet B (UVB) exposure. Vitamin D is essential for the maintenance of optimal bone and musculoskeletal health. It has also been suggested to play a role in the prevention of illness incidence, such as in upper respiratory tract infections (URTI). More recent research has indicated that an improved Vitamin D status may also play a role in enhancing exercise performance. Therefore, having a poor vitamin D status could negatively impact athletic training and competition. The purpose of this study is to evaluate the prevalence of vitamin D deficiency in university athletes and inactive controls in spring and autumn.

During this study the subjects will be asked to visit the labs on two occasions, at the beginning of the study for baseline measurements, and again on two occasions at the end of the study. Participants will have the following outcomes assessed: Sport performance (vertical jump height, muscular strength and aerobic fitness), peripheral Quantitative Computed Tomography (pQCT) scan of the bone mineral composition of the tibia, total body composition via Dual Energy X-ray Absorptiometry (DEXA),total and hip/femoral head bone mineral density and content to assess fracture risk via DEXA. Serum 25(OH)D levels (≈15ml of whole blood will be collected for these measurements. Dietary intake using self-reported food diaries. In addition illness and injury incidence will be recorded daily throughout the study in a booklet provided to the participants.Throughout the trial, the participants will be contacted via telephone/ email on a monthly basis to discuss any issues and maintain good communication.

DETAILED DESCRIPTION:
During this study the subjects will be asked to visit the labs on 4 different occasions. There will be two occasions, at the beginning of the study for baseline measurements, and again on two occasions at the end of the study.

Data collection will take place across two testing sessions (separated by ~24 - 72 hrs) in the Autumn and Spring period.

Session 1

* Peripheral Quantitative Computed Tomography (pQCT) scan of the bone mineral composition of the tibia.
* Total and percentage lean and fat mass and total bone mineral density via Dual Energy X-ray Absorptiometry (DEXA).
* Sport performance: Vertical jump height and maximal oxygen uptake (VO2 max) test.

Session 2

* Fasting serum 25(OH)D levels, lipid profile, glucose, insulin, serum calcium, albumin, parathyroid hormone, C- terminal telopeptide (CTX), full blood count, kidney, thyroid and liver function (≈15ml of whole blood will be collected for these measurements).
* Collection of self-reported food diaries to assess dietary intake
* Sport performance: muscular strength

Aerobic fitness will be tested using a VO2 max exercise protocol using a stationary cycle ergometer, the participants will be expected to perform this to maximal effort or exhaustion. The test will consist of progressive increments in cycling workload (power output, W) until volitional fatigue. The test will take about 8 - 12 minutes to complete and is dependent upon the fitness of the participants. This will take place in the Sport & Exercise Science laboratories based in the Clinical Investigation Unit (22AX00). All subjects will be supervised during exercise at all times and will implement an adequate warm-up and cool-down to minimize the risk of injury. Staff will be on hand throughout the testing trained adequately in basic life support (including defibrillation).

Muscular strength assessments will be performed at the Surrey Human Performance Institute. Muscular strength of the knee extensor and handgrip muscles will be determined using an Isokinetic Dynamometer and a handgrip dynamometer respectively. For each assessment three maximal effort isometric contractions will be performed and peak torque (nM) and strength (kg) will be recorded. Muscular power will be assessed through performance of a countermovement jump (CMJ).

Body composition (absolute and relative amount of lean and fat mass), whole body bone mineral density and hip and femur bone mineral density will be measured with the use of DEXA (located in the Sport & Exercise Science laboratories based in the Clinical Investigation Unit). Two scans will be performed: one for the assessment of whole body bone mineral density and body composition, and the other scan is performed to specifically assess fracture risk by scanning the hip and femoral head. Effective exposure doses for these scans are ~8uSv and ~4uSv respectively. The total effective dose is depending on the size ('thickness' & height) of the volunteer and is approximately equivalent to the cosmic radiation exposure received in 45min of a transatlantic flight, or the radiation dose received on eating 80g of Brazil nuts (Health Protection Agency).

Bone mineral content of the tibia will be assessed using pQCT and this will be correlated to bone mineral density data obtained from DEXA. One scan will be performed and effective exposure doses will be between 1.5-1.8uSv which is comparable to 10 min on a transatlantic flight or one handful of Brazil nuts. The estimated total exposure dose for a single subject during the entire study is ~28uSv which is the same level of exposure as an average UK citizen is exposed to over the course of 4 days via background radiation.

Results of the body composition, bone mineral density, jump height, muscular strength, aerobic fitness (maximal oxygen uptake: VO2max) and dietary intake from the self-reported food diaries will be made available to the subjects upon request. The results from the blood analysis will be reported to the subject if there are any health concerns raised. If the results are within healthy ranges the participants will not be contacted unless specifically requested for this information. The investigators will not be contacting their GPs if there are any concerns raised in the study however it will be stressed that participants should contact a GP to discuss the results found.

Upon commencing the study, the participants will be required to track their incidence of illness and training habits during the 20-week experimental period between baseline and conclusion measurements. Throughout this period the incidence of illness and days trained during the months must be recorded in a check-list booklet, which will be provided. An email reminder will be sent to prompt all participants to complete these booklets on a daily basis during the experimental period, this should only take 1-2 minutes every evening. Throughout the duration of the trial, the participants will be contacted via telephone/ email on a monthly basis to discuss any issues and maintain good communication.

ELIGIBILITY:
Inclusion Criteria:

University athlete inclusion criteria:

* Male or female
* Aged 18-30
* Regularly train/compete for Team Surrey Basketball, Boat Club, Swimming and Waterpolo, Netball or Rugby (for more than 4 hours/week)
* In good physical health
* Have a BMI >18 kg/m2
* Able to provide written informed consent

Control group inclusion criteria:

* Male or Female
* Age 18-30
* Do not use sun beds/ will not be going on a sun holiday/ returning home to a traditional sun holiday location between February 2017 and October 2017. This is because the results will be used to represent the Vitamin D status of young sporting individuals residing within the UK during these seasons.
* Do not take supplements containing Vitamin D
* Do not compete for Team Surrey and exercise less than 150 minutes / week.
* BMI: 18 - 30 kg/m2

Exclusion Criteria:

* Currently receiving treatment for medical conditions that are likely to affect vitamin D metabolism
* Hypercalcaemia (>2.5mmol/L)
* Regular use of sun-beds
* Having a sun holiday one month prior to commencing the study or plans for a sun holiday within the study period or will be returning home to a sun holiday location.
* Use of vitamin supplements containing vitamin D (if the prospective participants agrees to stop Vitamin D supplementation to join the study, a wash-out period of 8 weeks prior to commencing the trial would be acceptable).
* Excess alcohol intake for participants aged 18 years (> 21 units for males, > 14 units for females per week, as per Government guidelines)
* Those under dietary restriction (except vegetarianism) or following a weight-reducing diet.
* Clinically significant haematological abnormalities other than mild anaemia (Hb <12.0g/dl)
* Active malignancy
* Pregnant or planning a pregnancy during the study period

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the university population in Surrey during term-time
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Seasonal Change in the Number of Participants with Deficiency in Vitamin D (according to government cut-off points in the UK and USA) in University Athletes and their Healthy Controls. | 1 year
  This will be assessed by measuring serum 25(OH)D levels in participants during Autumn and Spring. Vitamin D status will be measured in nmol/L

SECONDARY OUTCOMES:
Seasonal Change in the Incidence of Injury in University Athletes | 1 year
  Self reported questionnaire
Seasonal Change in Bone Mineral Density in University Athletes | 1 year
  mg/cm
Seasonal Change in Bone Mineral Content in University Athletes | 1 year
  mg/cm
The change in vitamin D status due to participation in indoor or outdoor training in university level athletes between Autumn and Spring. | 1 year
  hours and nmol/L
Change between autumn and spring and the effects of high, medium and low impact sports on bone mineral density in university athletes | 1 year
  mg/cm
Changes from baseline in muscular power throughout an academic sporting season | 1 year
  Vertical jump: cm
Changes from baseline in muscular strength throughout an academic sporting season | 1 year
  hand-grip strength: kg, knee extensor muscular strength: nM
Changes from baseline in aerobic fitness throughout an academic sporting season | 1 year
  ml/kg/min-1
Change from baseline in the incidence of injury and illness and its correlation with vitamin D status | 1 year
  Days of illness reported or missed training due to injury

CONTACTS AND LOCATIONS:
Overall Officials: Susan Lanham-New, Ph.D, Study Chair — Head, Department of Nutritional Scienes
Locations (2):
- United Kingdom (2):
  - Surrey Human Performance Institute, Guildford, Surrey
  - University of Surrey, Guildford, Surrey

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Halliday TM, Peterson NJ, Thomas JJ, Kleppinger K, Hollis BW, Larson-Meyer DE. Vitamin D status relative to diet, lifestyle, injury, and illness in college athletes. Med Sci Sports Exerc. 2011 Feb;43(2):335-43. doi: 10.1249/MSS.0b013e3181eb9d4d. PMID 20543748
- [Background] Close GL, Leckey J, Patterson M, Bradley W, Owens DJ, Fraser WD, Morton JP. The effects of vitamin D(3) supplementation on serum total 25[OH]D concentration and physical performance: a randomised dose-response study. Br J Sports Med. 2013 Jul;47(11):692-6. doi: 10.1136/bjsports-2012-091735. Epub 2013 Feb 14. PMID 23410885
- [Background] Farrokhyar F, Tabasinejad R, Dao D, Peterson D, Ayeni OR, Hadioonzadeh R, Bhandari M. Prevalence of vitamin D inadequacy in athletes: a systematic-review and meta-analysis. Sports Med. 2015 Mar;45(3):365-78. doi: 10.1007/s40279-014-0267-6. PMID 25277808

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT03253055/Prot_SAP_000.pdf